CLINICAL TRIAL: NCT06913491
Title: Efficacy of PEEK Acuity Versus ETDRS Chart for Assessment of Visual Acuity and Refractive Error
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/803
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Visual acuity is a key indicator of visual function, often measured using the ETDRS chart, the gold standard in clinical settings. However, the increasing need for accessible and cost-effective screening tools, especially in underserved areas, has led to the development of mobile health applications like the Peek Acuity application.

DETAILED DESCRIPTION:
This study aims to compare the diagnostic accuracy and efficiency of the Peek acuity application (Portable Eye Examination Kit) with the ETDRS (Early Treatment of Diabetic Retinopathy Study) chart in assessing visual acuity and refractive errors. The study will involve 58 participants, selected using a non-probability convenience sampling technique. A comparative cross-sectional design will be used.

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* 18 years of age or older.
* Individuals with normal vision or those with refractive error who had their corrected glasses.
* Individuals who are willing and able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Individuals with anterior segment abnormalities such as conjunctivitis, Iritis, uveitis, keratitis, or corneal ulcers.
* Individuals with vision deprivation due to corneal opacities, cataracts, glaucoma, retinal, and optic nerve pathologies.
* Postoperative/intraoperative complications.
* Have received mydriatic drops.
* Individuals who cannot achieve normal visual acuity with corrective lenses (glasses or contact lenses).
* Individuals with neurological conditions affecting vision
* Individuals unable to cooperate with visual acuity testing due to cognitive impairments or language barriers.
* Individuals who have had refractive surgery or other eye treatments within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Visual acuity is a key indicator of visual function, often measured using the ETDRS chart, the gold standard in clinical settings. However, the increasing need for accessible and cost-effective screening tools, especially in underserved areas,
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Peek Acuity | 12 Months
  Peek Acuity is easier to administer than an equivalent wall chart, such as Snellen or ETDRS, and is generally quicker to complete. The algorithm that controls progress through each test is optimised for clinical accuracy, so the test will end just as soon as a reliable score has been obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Eagle Eyes Relief Trust FF120, Divine mega 2, new airport road, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No